CLINICAL TRIAL: NCT02034656
Title: Patterns of ABL Mutation in Asian With Imatinib Resistant Chronic Myeloid Leukemia and Ph Positive Acute Lymphocytc Leuekmia Patients (AMICA): A Retrospective Feasibility Study
Brief Title: Patterns of ABL Mutation in Asian With Imatinib Resistant Chronic Myeloid Leukemia and Ph Positive Acute Lymphocytc Leuekmia Patients (AMICA)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Dong-Wook Kim, Professor, Seoul St. Mary's Hospital
Other Study IDs: KC10RSGI0437
Record Dates: First submitted 2012-07-27; First posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Myeloid Leukemia or Ph Positive ALL
Keywords: imatinib resistance; mutation
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- imatinib resistance: All mutation data from CML and Ph positive ALL patients who developed imatinib resistance during the year 2001-2009

SUMMARY:
The purposes of this study are to investigate the patterns of BCR-ABL mutations in CML and Ph positive ALL patients with imatinib resistance during the year of 2001-2009 in Asian institutes.

DETAILED DESCRIPTION:
Awareness of the significance of BCR-ABL mutations is generally low across Asia. This is partly due to historical limitations in capabilities for mutation testing. While numerous mutation studies have been done in non-Asian populations, there are very few published reports on mutations in Asians. CML management in Asia therefore continues to be largely intuitive.

Anecdotal reports, suggest that there may differences in the presence or absence of mutations at the time of initial diagnosis and their occurrence during imatinib treatment. At present, however, we have no comprehensive formal knowledge of the actual nature of mutations in Asians. There are moves towards the establishment of CML registries that will capture the pattern of mutations among Asian patients.

In recent years, several laboratories in the region have been performing mutation analysis. However, no systematic evaluation of or report on these data has been undertaken. This study therefore intends to collect documented mutation data in Asian CML and Ph positive ALL patients from identified Asian institutes. While this is a retrospective, cross-sectional analysis of mutation information, the study will provide the first comprehensive formal report on mutations in Asian CML and Ph positive ALL patients. The collecting information has the potential better to inform the clinical management of CML and Ph positive ALL in Asia according to the mutation result and possibly future research in these patients.

ELIGIBILITY:
Inclusion Criteria:

* All mutation data from CML and Ph positive ALL patients who developed imatinib resistance during the year 2001-2009

Exclusion Criteria:

* Mutation data from CML and Ph positive ALL patients who, in addition to imatinib, received other therapy. Follow up mutation report after second generation TKI therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean Adult CML or Ph positive ALL patients
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2010-07; Primary Completion 2014-03 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Analyzing the patterns and rate of BCR-ABL mutations in Asian CML and Ph positive ALL patients | 9 years
  To describe the patterns and rate of BCR-ABL mutations in Asian CML and Ph positive ALL patients. To compare the patterns of BCR-ABL mutations to that of Non-Asian. To describe methods used in mutation analysis

SECONDARY OUTCOMES:
Description of the choice of second-line therapy | 9 years
  To describe about the choice of second-line therapy To describe outcome after emergence of resistance according to type of mutation

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Wook Kim, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea